CLINICAL TRIAL: NCT05101408
Title: Combining Executive Training and Anomia Therapy in Chronic Post-stroke Aphasia : a Single Case Experimental Design -SCED Preliminary Study
Brief Title: Executive Training and Anomia Therapy in Chronic Post-stroke Aphasia
Acronym: ETAT PSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0597
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Anomia; Post-stroke Aphasia
Keywords: Aphasia; Speech-Language Therapy; Anomia; Executive functions
MeSH Terms: conditions — Anomia; Aphasia; Communication Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aphasia is a devastating acquired language impairment mainly caused by stroke, in which anomia is a quintessential clinical feature. If speech-language therapy (SLT) has been shown to be effective for persons with aphasia, the relative efficiency of one SLT strategy over another remains a matter of debate. The influential relationship between language, executive functions and aphasia rehabilitation outcomes has been addressed in a number of studies, but only few of them have studied the effect of adding an executive training to linguistic therapies.The aim of this study is to measure the efficiency of a protocol combining anomia therapy and executive training on naming skills and discourse in post-stroke aphasic persons at the chronic stage

ELIGIBILITY:
Inclusion criteria:

* 18 < age > 80 years
* adult person with chronic post-stroke aphasia (> 6 months postonset)
* receiving SLT rehabilitation 3 times a Week

Exclusion criteria:

* presence of apraxia of speech
* major impairment of comprehension
* history of other neurological or psychiatric disease

Exclusion criteria:

* presence of apraxia of speech
* presence of major impairment of comprehension
* presence of history of other neurological or psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Person with post-stroke aphasia at the chronic stage, receiving SLT rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Evolution of individual naming scores | 2 days
  Evolution of individual naming scores during baseline and treatment phases Participants are asked to name pictures from a personal naming task constituted of 100 black and white pictures and scores are expressed as percent of correct responses (min 0, max 100): higher percents meaning a better outcome. A visual analysis of the evolution of these scores along the course of the treatment will be conducted.
Comparison of discourse | 2 days
  Comparison of discourse scores before and after the treatment For each participant, four different samples of discourse are elicited before and after the treatment (picture description, personal narrative, book supported narrative, procedural information). The mean number of correct words per minute is then computed for each participant, and compared between the two time points, higher scores meaning a better outcome.

SECONDARY OUTCOMES:
Comparison of executive scores | 2 days
  Comparison of executive scores before and after the treatment Executive scores are computed before and after treatment for each participant, from the Modified Card Sorting Test (Nelson, 1976), in which higher number of categories achieved means a better outcome, and from a verbal fluency task in which higher number of words produced in 2 minutes means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Moritz-Gasser, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC